CLINICAL TRIAL: NCT03029364
Title: Body Composition and Lipid Metabolism at Rest and During Exercise: A Cross-Sectional Analysis.
Status: Completed | Type: Observational
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Lecturer (Assistant Professor) in Human Physiology, University of Bath
Other Study IDs: 17/SW/0269
Record Dates: First submitted 2017-01-14; First posted 2017-01-24 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Lipid Metabolism; Substrate Metabolism; Exercise
Keywords: Maximal Fat Oxidation; Exercise; Intra-individual variability; Determinants; Whole-body fat oxidation; Body composition
MeSH Terms: conditions — Motor Activity | interventions — Clinical Protocols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum and buffy coat layer extraction from blood samples. Skeletal muscle and adipose tissue (fat) samples. Urine sample for immediate analysis and disposal.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Male and Female Adults: Completion of Study Protocol
  Interventions: Behavioral: Study Protocol

INTERVENTIONS:
Behavioral: Study Protocol — Participants will complete three study protocols 7 - 28 days apart which includes:
  * 3 x main trial days (max. 150 mins) involving body composition analysis, indirect calorimetry, a blood sample, optional muscle and / or adipose tissue biopsies and a maximal cardiorespiratory fitness test.
  * 2 x lifestyle monitoring periods (physical activity and diet) for the prior 7 days before each main trial day.
  * Maintenance of habitual habits, dietary and physical activity behaviour patterns
  We are observing biological / health parameters in a group of individuals who will be assessed under resting and exercising conditions. The current study does not involve an intervention.

SUMMARY:
The ability to upregulate fat oxidation at appropriate times such as during fasting, low to moderate intensity exercise and after a high fat meal, is popularly advocated. This is presumably due to the perception that a high capacity to utilise fat may improve (ultra) endurance performance and help in the regulation of body fat and metabolic diseases. In accordance, impaired fat use at rest has been associated with obesity and insulin resistance (Kelley et al., 1999). However, there is inconclusive and / or a lack of systematic evidence, especially in a large diverse range of adults, exploring:

1) Whether whole body fat use during exercise is altered in individuals with overweight or obesity compared to lean individuals

3) The intra-individual variability in whole-body fat use at rest and during exercise

4) Physiological, metabolic, lifestyle and genetic characteristics that are associated with whole-body fat use at rest and during exercise

Therefore, the objectives of this study are three-fold:

1. To explore whether whole body fat use is associated with body composition
2. To explore associations between whole-body fat use and physiological, metabolic, lifestyle and genetic variables
3. To assess the intra-individual variability of whole-body fat use.

This study is an observational, exploratory cross-sectional study. A wide range of 'healthy' and 'at-risk of metabolic disease' adults will be recruited.

Participants will be asked to visit a laboratory at the University of Bath four times. Visit 1 is a screening and study familiarisation visit. Visits 2 and 3 are to be completed within 7-14 days and involve lifestyle monitoring (dietary and physical activity), a one-off urine and blood sample, assessment of fuel use at rest and during exercise (the latter through an incremental graded cycling exercise test to exhaustion). Visit 4 is to assess body composition via a dual-energy x-ray absorptiometry (DEXA) scan in addition to an optional skeletal muscle and / or fat tissue biopsy.

DETAILED DESCRIPTION:
Metabolic flexibility broadly refers to the ability to utilize the right fuel source for energy (primarily either carbohydrate or fat) at the right time (Kelley and Mandarino, 2000). This was first conceptualised at the level of skeletal muscle (Kelley and Mandarino, 1990; Andres et al., 1956). A main tenant originally captured by 'metabolic flexibility' is the predominant utilization of fat as an energy source under rested post-absorptive conditions in 'healthy' individuals (Kelley et al., 1999; Kelley and Mandarino, 1990). Recently, there has been a call to extend the concept of 'metabolic flexibility' to exercising conditions (Goodpaster and Sparks, 2017; Rynders et al., 2017). Similarly to at rest, fat provides an important source of energy during low-to-moderate intensity exercise (van Loon et al., 2001; Romijn et al., 1993). Thus, in healthy individuals at the whole-body and skeletal muscle level, it is robustly characterised and accepted that fat is an important and predominant fuel source for energy under such conditions.

However, it is commonly proposed that a lower reliance upon fat as a fuel source is present in individuals with obesity and type 2 diabetes and consequently, has been implicated in the pathogenesis of such conditions (Rynders et al., 2017; Kelley and Mandarino, 2000). Alternatively, a high capacity to utilize fat under the aforementioned two situations is advocated to be a desirable trait for both athletes and non-athletes, presumably due to the perception that high rates of fat utilization may improve endurance performance and/or assist with the regulation of body fat and metabolic health. As such, much interest has been generated into upregulating fat utilization at appropriate times e.g. during fasting and low-to-moderate intensity exercise.

Correspondingly, lower resting and exercising fat use has been reported in individuals with obesity vs lean (e.g. Lanzi et al., 2014; Perez-Martin et al., 2001; Kelley et al., 1999). Furthermore, greater fat use at rest has been associated with lower future body weight and fat gain / regain (e.g. Shook et al., 2016; Seidell et al., 1992), and during exercise with reduced short term post-exercise energy intake / balance (e.g. Hopkins et al., 2012), exercise-induced fat loss (Barwell et al., 2008) and weight loss / maintenance (Dandadell et al., 2017). Importantly, however, this relationship is not always apparent with similar (e.g. Blaize et a., 2014; Croci et al., 2014) or higher (e.g. Ara et al., 2011; Goodpaster et al., 2002; Horowtiz et al., 2000) rates of fat use at rest and during exercise reported in individuals with obesity compared to lean counterparts. Furthermore, cross-sectional and prospective associations do not always exist between lower fat use and greater body weight / fat mass gain or regain (e.g. Dandanell et al., 2017; Ellis et al., 2010). Thus, despite being popularly advocated, it is currently unclear whether lower fat use at rest or during exercise predisposes or is a characteristic of excess adiposity (i.e. obesity).

The inconsistent findings could partly be due to numerous methodological discrepancies between studies such as participant characteristics, matching of comparative groups, the exercise protocol utilised and / or the assessment of body composition, lipid oxidation and cardio-respiratory fitness levels.

Therefore, through the use of well-established and respected techniques, we aim to comprehensively and systematically explore whether whole-body fat use at rest and during exercise is:

1. Altered in individuals with overweight or obesity compared to lean individuals
2. Further determinants / factors that may influence fat use
3. The intra-individual variation in fat use which will help to more confidently determine the above objectives.

ELIGIBILITY:
Inclusion Criteria:

* be between 18 - 65 years of age
* male or female
* body mass index between 18.9 - 35 kg/m2
* be able and willing to give informed oral and written consent
* complete and meet the defined criteria of pre-study questionnaires and screens

Exclusion Criteria:

* Currently have or have a previous history of metabolic, cardio-pulmonary or musculoskeletal disease
* BMI below 18.9 or above 35 kg/m2
* Have plans to change lifestyle (diet and/or physical activity) during the study period ( 7 - 21 days)
* Unwillingness or unable to sufficiently meet study demands

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Maximal rate of whole-body fat oxidation (mg/kg FFM/min) | 7 - 14 days
  Fat free mass (FFM). Assessed during the incremental stage maximal cardio-respiratory fitness test

SECONDARY OUTCOMES:
Maximal rate of whole-body fat oxidation (g/min) | 7-14 days
  Non-adjusted rate. Assessed during the incremental stage maximal cardio-respiratory fitness test
FATmax (% of maximum oxygen consumption) | 7 - 14 days
  The exercise intensity that maximal rate of whole-body fat oxidation occurs at. Expressed as % of VO2peak). Assessed during the incremental stage maximal cardio-respiratory fitness test.
FATmax (% of Watt max) | 7 - 14 days
  The exercise intensity that maximal rate of whole-body fat oxidation occurs at. Expressed as % of Watt max). Assessed during the incremental stage maximal cardio-respiratory fitness test.
FATmax (% of Heart Rate max) | 7 - 14 days
  The exercise intensity that maximal rate of whole-body fat oxidation occurs at. expressed either as % of heart rate max). Assessed during the incremental stage maximal cardio-respiratory fitness test
Whole-body substrate oxidation rates (Carbohydrates and Lipid) during exercise | 7 - 14 days
  Assessed during the incremental stage maximal cardio-respiratory fitness test via indirect calorimetry of expired gas samples.
Whole-body substrate oxidation rates (Carbohydrates and Lipid) at rest | 7 - 14 days
  Assessed at rest through the participant lying in a semi-supine position via indirect calorimetry of expired gas samples.
Resting metabolic rate | 7 - 14 days
  Assessed at rest through the participant lying in a semi-supine position via indirect calorimetry of expired gas samples.
Cardiorespiratory fitness (VO2peak) | 7 - 14 days
  Assessed during the incremental stage maximal cardio-respiratory fitness test
Habitual Energy Intake | 7 - 21 days
  Participants will be asked to complete a self-weighed food and drink diary before each main trial day (Visit 2 and 3) so that average daily calorie and macronutrient intake can be calculated. The procedure will be explained by the CI. This diet monitoring period must include 3 week-days, at least one 1 weekend day and the immediate 48-hrs prior to the beginning of each main trial (Visit 2 and 3). Additionally, the prior 48-hrs before Visit 2 will be replicated before Visit 3.
Habitual Energy Expenditure / Physical Activity | 7 - 21 days
  Physical activity will be measured by accelerometry and heart-rate monitoring for 7 days before each main trial day (Visit 2 and 3). This procedure will be explained by the CI. ntake can be calculated. The participants physical activity levels for the immediate 48-hrs prior to the beginning of each main trial (Visit 2 and 3) will be asked to be replicated as closely as possible.
Menstrual Cycle (females only) | 7 - 21 days
  Assessed through a self-reported menstrual cycle questionnaire
Self-reported Physical Activity level | 7-21 days
  Assessed by the International Physical Activity Questionnaire (long form)
Fasting glucose concentration | 7-21 days
  Assessed via plasma sample extracted from the blood sample
Fasting lipid profiles (triglycerides / cholesterol) | 7-21 days
  Assessed via serum sample extracted from the blood sample
Fasting Adipose tissue derived hormone concentrations (leptin, adiponectin) | 7-21 days
  Assessed via plasma sample extracted from the blood sample
Fasting catecholamine concentrations (epinephrine and norepinephrine) | 7-21 days
  Assessed via plasma sample extracted from the blood sample
Fasting sex hormone concentrations (17 beta-estradiol, testosterone, progesterone) | 7-21 days
  Assessed via serum sample extracted from the blood sample
Fasting pancreatic derived hormone concentrations (insulin and glucagon) | 7-21 days
  Assessed via plasma sample extracted from the blood sample
Hydration Status (urine specific gravity) | 7-21 days
  Assessed via analysis of urine sample with a refractometer
Age | 7-21 days
  Assessed via a participant questionnaire
Sex | 7-21 days
  Assessed via a participant questionnaire
Ethnicity | 7-21 days
  Assessed via a participant questionnaire
Smoking Status | 7-21 days
  Assessed via a participant questionnaire
Medication / supplement use | 7-21 days
  Assessed via a participant questionnaire
Dietary pattern / requirements (e.g. vegetarian, vegan, Celiac disease) | 7-21 days
  Assessed via a participant questionnaire
Body Mass (kg) | 7-21 days
  Assessed via body weighing scales
Body Mass Index (kg/m2) | 7-21 days
  Assessed by dividing body weight in kg by height in metres squared.
Waist circumference (cm) | 7-21 days
  Assessed via use of an anthropometric tape measure
Hip Circumference (cm) | 7-21 days
  Assessed via use of an anthropometric tape measure
Body fat percentage | 1 day
  Assessed via a dual energy xray absorptiometry scan at Visit 4.
Body fat localisation | 1 day
  Assessed via a dual energy xray absorptiometry scan at Visit 4.
Lean body mass | 1 day
  Assessed via a dual energy xray absorptiometry scan at Visit 4.
Body fat percentage | 7-21 days
  Bioelectrical Impedance Analysis from the body weighing scales
Genotyping analysis | 7 - 21 days
  Genotyping analysis will be assessed through the extraction of the buffy coat layer from the blood sample
Skeletal Muscle sample (Optional) | 1 day
  The optional muscle sample will be obtained from the quadriceps muscle using the Bergstrom technique on Visit 4.
Adipose Tissue (Fat) sample (Optional) | 1 day
  The optional fat sample will be obtained from the subcutaneous abdominal region (5 cm laterally of the umbilicus) via the 'lipoaspiration' technique on Visit 4.
Fat mass index (body fat in kg/m2) | 7 - 21 days
  Assessed by dividing body fat in kg by height in metres squared.

CONTACTS AND LOCATIONS:
Overall Officials: Javier T Gonzalez, PhD, Principal Investigator — University of Bath
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kelley DE, Mandarino LJ. Fuel selection in human skeletal muscle in insulin resistance: a reexamination. Diabetes. 2000 May;49(5):677-83. doi: 10.2337/diabetes.49.5.677. PMID 10905472
- [Background] Kelley DE, Mandarino LJ. Hyperglycemia normalizes insulin-stimulated skeletal muscle glucose oxidation and storage in noninsulin-dependent diabetes mellitus. J Clin Invest. 1990 Dec;86(6):1999-2007. doi: 10.1172/JCI114935. PMID 2123890
- [Background] ANDRES R, CADER G, ZIERLER KL. The quantitatively minor role of carbohydrate in oxidative metabolism by skeletal muscle in intact man in the basal state; measurements of oxygen and glucose uptake and carbon dioxide and lactate production in the forearm. J Clin Invest. 1956 Jun;35(6):671-82. doi: 10.1172/JCI103324. No abstract available. PMID 13319506
- [Background] Goodpaster BH, Sparks LM. Metabolic Flexibility in Health and Disease. Cell Metab. 2017 May 2;25(5):1027-1036. doi: 10.1016/j.cmet.2017.04.015. PMID 28467922
- [Background] Rynders CA, Blanc S, DeJong N, Bessesen DH, Bergouignan A. Sedentary behaviour is a key determinant of metabolic inflexibility. J Physiol. 2018 Apr 15;596(8):1319-1330. doi: 10.1113/JP273282. Epub 2017 Jul 4. PMID 28543022
- [Background] van Loon LJ, Greenhaff PL, Constantin-Teodosiu D, Saris WH, Wagenmakers AJ. The effects of increasing exercise intensity on muscle fuel utilisation in humans. J Physiol. 2001 Oct 1;536(Pt 1):295-304. doi: 10.1111/j.1469-7793.2001.00295.x. PMID 11579177
- [Background] Romijn JA, Coyle EF, Sidossis LS, Gastaldelli A, Horowitz JF, Endert E, Wolfe RR. Regulation of endogenous fat and carbohydrate metabolism in relation to exercise intensity and duration. Am J Physiol. 1993 Sep;265(3 Pt 1):E380-91. doi: 10.1152/ajpendo.1993.265.3.E380. PMID 8214047
- [Background] Lanzi S, Codecasa F, Cornacchia M, Maestrini S, Salvadori A, Brunani A, Malatesta D. Fat oxidation, hormonal and plasma metabolite kinetics during a submaximal incremental test in lean and obese adults. PLoS One. 2014 Feb 11;9(2):e88707. doi: 10.1371/journal.pone.0088707. eCollection 2014. PMID 24523934
- [Background] Perez-Martin A, Dumortier M, Raynaud E, Brun JF, Fedou C, Bringer J, Mercier J. Balance of substrate oxidation during submaximal exercise in lean and obese people. Diabetes Metab. 2001 Sep;27(4 Pt 1):466-74. PMID 11547220
- [Background] Kelley DE, Goodpaster B, Wing RR, Simoneau JA. Skeletal muscle fatty acid metabolism in association with insulin resistance, obesity, and weight loss. Am J Physiol. 1999 Dec;277(6):E1130-41. doi: 10.1152/ajpendo.1999.277.6.E1130. PMID 10600804
- [Background] Shook RP, Hand GA, Paluch AE, Wang X, Moran R, Hebert JR, Jakicic JM, Blair SN. High respiratory quotient is associated with increases in body weight and fat mass in young adults. Eur J Clin Nutr. 2016 Oct;70(10):1197-1202. doi: 10.1038/ejcn.2015.198. Epub 2015 Nov 25. PMID 26603877
- [Background] Seidell JC, Muller DC, Sorkin JD, Andres R. Fasting respiratory exchange ratio and resting metabolic rate as predictors of weight gain: the Baltimore Longitudinal Study on Aging. Int J Obes Relat Metab Disord. 1992 Sep;16(9):667-74. PMID 1328091
- [Background] Hopkins M, Blundell JE, King NA. Individual variability in compensatory eating following acute exercise in overweight and obese women. Br J Sports Med. 2014 Oct;48(20):1472-6. doi: 10.1136/bjsports-2012-091721. Epub 2013 May 10. PMID 23666018
- [Background] Barwell ND, Malkova D, Leggate M, Gill JM. Individual responsiveness to exercise-induced fat loss is associated with change in resting substrate utilization. Metabolism. 2009 Sep;58(9):1320-8. doi: 10.1016/j.metabol.2009.04.016. Epub 2009 Jun 18. PMID 19501861
- [Background] Dandanell S, Husted K, Amdisen S, Vigelso A, Dela F, Larsen S, Helge JW. Influence of maximal fat oxidation on long-term weight loss maintenance in humans. J Appl Physiol (1985). 2017 Jul 1;123(1):267-274. doi: 10.1152/japplphysiol.00270.2017. Epub 2017 May 25. PMID 28546468
- [Background] Blaize AN, Potteiger JA, Claytor RP, Noe DA. Body fat has no effect on the maximal fat oxidation rate in young, normal, and overweight women. J Strength Cond Res. 2014 Aug;28(8):2121-6. doi: 10.1519/JSC.0000000000000512. PMID 24796985
- [Background] Croci I, Hickman IJ, Wood RE, Borrani F, Macdonald GA, Byrne NM. Fat oxidation over a range of exercise intensities: fitness versus fatness. Appl Physiol Nutr Metab. 2014 Dec;39(12):1352-9. doi: 10.1139/apnm-2014-0144. Epub 2014 Aug 1. PMID 25356842
- [Background] Ara I, Larsen S, Stallknecht B, Guerra B, Morales-Alamo D, Andersen JL, Ponce-Gonzalez JG, Guadalupe-Grau A, Galbo H, Calbet JA, Helge JW. Normal mitochondrial function and increased fat oxidation capacity in leg and arm muscles in obese humans. Int J Obes (Lond). 2011 Jan;35(1):99-108. doi: 10.1038/ijo.2010.123. Epub 2010 Jun 15. PMID 20548301
- [Background] Horowitz JF, Klein S. Oxidation of nonplasma fatty acids during exercise is increased in women with abdominal obesity. J Appl Physiol (1985). 2000 Dec;89(6):2276-82. doi: 10.1152/jappl.2000.89.6.2276. PMID 11090579
- [Background] Goodpaster BH, Wolfe RR, Kelley DE. Effects of obesity on substrate utilization during exercise. Obes Res. 2002 Jul;10(7):575-84. doi: 10.1038/oby.2002.78. PMID 12105277
- [Background] Ellis AC, Hyatt TC, Hunter GR, Gower BA. Respiratory quotient predicts fat mass gain in premenopausal women. Obesity (Silver Spring). 2010 Dec;18(12):2255-9. doi: 10.1038/oby.2010.96. Epub 2010 May 6. PMID 20448540

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03029364/Prot_SAP_001.pdf